CLINICAL TRIAL: NCT06743139
Title: Evaluation of Effort Limitation Parameters of Patients With Homozygous Sickle Cell Disease
Brief Title: Exploration of the Parameters Influencing the Effort Limitation of Patients Suffering From Homozygous Sickle Cell Anemia
Acronym: PHYSIO-EXDRE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201322
Record Dates: First submitted 2022-06-27; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-07

CONDITIONS: Analyze the Results of Cardiorespiratory Stress Tests; Resting and Stress Echocardiography; Capillary Lactatemia Measurements at the Ear
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echography — Simultaneous performance of an echocardiogram (part of the follow-up assessment for sickle cell heart disease) at rest and then during the cardiorespiratory stress test, and an ear capillary lactatemia analysis (already routinely performed to ensure the safety of the cardiorespiratory stress test) during the cardiorespiratory stress test routinely performed at Mondor University Hospital prior to cardiovascular rehabilitation programs.

SUMMARY:
The cardiovascular complications of sickle cell disease are associated with major morbidity and mortality, as well as impaired quality of life. Stratifying the cardiovascular risk of these patients solely on resting parameters (blood pressure, cardiac ultrasound) is limited. The hypothesis that an exhaustive analysis of the physiological parameters of exercise is launched allows more relevant phenotyping and therefore much better stratification of the individual risk of these patients..

Recent studies have shown a paradigm shift in the use of physical activity. Hitherto inadvisable (acidosis, vaso-occlusive crises), if adapted, moderate and regular, it can lead to functional improvement and a reduction in crises. As a result, cardiovascular exercise rehabilitation is becoming increasingly popular in this population.

It's easy to see how effort assessment, particularly through cardiorespiratory exchanges, will become more common in this pathology, making its analysis accessible and interesting.

DETAILED DESCRIPTION:
The cardiovascular complications of sickle cell disease are associated with major morbidity and mortality, as well as impaired quality of life. Stratifying the cardiovascular risk of these patients solely on resting parameters (blood pressure, cardiac ultrasound) is limited. The hypothesis that an exhaustive analysis of the physiological parameters of exercise is launched allows more relevant phenotyping and therefore much better stratification of the individual risk of these patients.

Recent studies have shown a paradigm shift in the use of physical activity. Hitherto inadvisable (acidosis, vaso-occlusive crises), if adapted, moderate and regular, it can lead to functional improvement and a reduction in crises. As a result, cardiovascular exercise rehabilitation is becoming increasingly popular in this population.

It's easy to see how effort assessment, particularly through cardiorespiratory exchanges, will become more common in this pathology, making its analysis accessible and interesting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years old
* Affiliated with a social security scheme (beneficiary or beneficiary's beneficiary)

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients under guardianship, curatorship or legal protection
* Patient under AME
* Patient with a contraindication or unsuitability for physical activity on a cycloergometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with homozygous sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
To define different clinico-biological profiles in patients with sickle cell disease (HbSS) | 4 weeks
  To define different clinico-biological profiles in patients with sickle cell disease (HbSS) by means of an exhaustive physiological analysis coupled with exercise.

SECONDARY OUTCOMES:
Study resting characteristics to identify at an early stage patients with potential cardiac alterations. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'HUMIERES, Dr, Study Director — Henri Mondor University Hospital
Locations (1):
- Assistance Publique Hôpitaux de Paris-Hôpital Henri Mondor, Créteil, Paris, France

IPD SHARING:
Plan to Share IPD: No
Les données sont la propriété de l'APHP

REFERENCES:
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] http://beh.santepubliquefrance.fr/beh/2015/8/2015_8_2.html
- [Background] Fitzhugh CD, Lauder N, Jonassaint JC, Telen MJ, Zhao X, Wright EC, Gilliam FR, De Castro LM. Cardiopulmonary complications leading to premature deaths in adult patients with sickle cell disease. Am J Hematol. 2010 Jan;85(1):36-40. doi: 10.1002/ajh.21569. PMID 20029950
- [Background] Hammoudi N, Lionnet F, Redheuil A, Montalescot G. Cardiovascular manifestations of sickle cell disease. Eur Heart J. 2020 Apr 1;41(13):1365-1373. doi: 10.1093/eurheartj/ehz217. PMID 31005979
- [Background] Guazzi M, Bandera F, Ozemek C, Systrom D, Arena R. Cardiopulmonary Exercise Testing: What Is its Value? J Am Coll Cardiol. 2017 Sep 26;70(13):1618-1636. doi: 10.1016/j.jacc.2017.08.012. PMID 28935040